CLINICAL TRIAL: NCT04464421
Title: Pilot Test of Contingency Management and Brief Motivational Interviewing + Substance Free Activity Session Interventions + Mindfulness-Based Adherence Promotion
Brief Title: SMART Effectiveness Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karen Derefinko, PhD (Other)
Collaborators: University of Memphis (Other); University of New Mexico (Other)
Responsible Party: Sponsor-Investigator, Karen Derefinko, PhD, Associate Professor, University of Tennessee
Organization: University of Tennessee (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-07418-XP UM
Record Dates: First submitted 2020-06-23; First posted 2020-07-09 (Actual); Results first posted 2022-09-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Opioid-use Disorder; Opioid Dependence; Treatment Adherence
Keywords: opioid use disorder; OUD; buprenorphine; treatment adherence; substance-free activities; brief motivational interviewing; contingency management
MeSH Terms: conditions — Opioid-Related Disorders; Treatment Adherence and Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency management (CM) (Experimental): Participants received incentives for urine toxicology with a positive result for Buprenorphine metabolites at each of the first four visits after initiation of Buprenorphine-Naloxone.
  Interventions: Behavioral: Contingency Management (CM)
- BSM (Experimental): BSM (Brief Motivational Intervention + Substance Free Activities Session + Mindfulness-Based Adherence Promotion) participants had one-on-one behavioral intervention sessions at each of the first four visits after initiation of Buprenorphine-Naloxone.
  Interventions: Behavioral: Brief Motivational Intervention + Substance Free Activities Session + Mindfulness-Based Adherence Promotion (BSM)

INTERVENTIONS:
Behavioral: Contingency Management (CM) — Participants were able to draw a gift card from a virtual fishbowl when their urine toxicology results are positive for buprenorphine metabolites. Gift card values were $25, $50, or $100.
  Arms: Contingency management (CM)
Behavioral: Brief Motivational Intervention + Substance Free Activities Session + Mindfulness-Based Adherence Promotion (BSM) — Participants had one-on-one sessions with a behavioral interventionist to discuss their goals regarding treatment, how to reach these goals, the importance of substance-free activities, and mindfulness skills.
  Arms: BSM

SUMMARY:
The current study piloted two psychosocial interventions developed to increase buprenorphine-naloxone adherence in individuals with opioid use disorder (OUD). Participants were randomized to receive either contingency management (CM) or a brief substance free activities session plus mindfulness (BSM) cognitive-behavioral intervention. Participants were 48 newly presenting patients from an OUD treatment clinic. The primary outcome was medication adherence, as measured by buprenorphine metabolite in urine and presence at 2 or more of 4 possible physician visits.

DETAILED DESCRIPTION:
We engaged with referred OUD patients at the time of their initial visit to the clinic. Interested patients were informed about the study in a private room, and if eligible, were consented and randomized to condition. Randomization occurred in blocks of 4. At the next physician visit, participants engaged in their first intervention activities (either CM or BSM). This was repeated for the following 3 physician visits.

CM. Contingency Management (CM). The CM intervention provided participants with a gift card at each of the first 4 follow up physician visits to the clinic where the participant's urine showed evidence of buprenorphine use. The strategy for CM rewards was based upon Petry's "fishbowl" draw, where variable values of gift cards were available for draw at each positive buprenorphine urine toxicology result. For the current study, which was conducted when COVID safety requirements were still high, a computerized "picker wheel" was used rather than an actual fishbowl to reduce possible viral transmission. Participants watched the wheel spin and told the interventionist when to stop the spin, at which time the value of the gift card was displayed. The picker wheel was programmed to include a 60% chance of a $25 gift card, a 20% chance of a $50 gift card, and a 20% chance of a $100 gift card. The average (expected) value of gift cards at this rate was $45 (or $180 total across 16 weeks, well below the typical range used in similar work).

BSM. Brief Motivational Interviewing plus Substance Free Activities Session plus Mindfulness (BSM). The BSM intervention included the following topics: (1) Short and Long-Term Goals: Identifying goals (e.g., What are your goals for this month…for the next 5 years?), requirements needed to achieve these goals (e.g., What would you need to do to achieve those goals?) and the potential role of relapse in jeopardizing these goals; (2) Personalized Feedback on Recent Time Allocation: (e.g., time spent with family, work, education/hobbies/creative activities, exercise/time in nature/self-care, watching tv/surfing the internet, religious or spiritual activities, recovery and nonrecovery activities; along with open ended questions asking about the extent to which their recent time allocation is consistent with their goals and values; (3) Episodic Future Thinking: An experiential intervention that prompts individuals to describe personal, emotional, and situational details of a valued future outcome that they desire; (4) Substance Free Activities: Based upon named hobbies and interests, participants were offered a personalized list of locally available substance-free activities developed by the interventionist; (5) Stop Observe Breathe Expand Respond (SOBER) Breathing Space: This exercise is intended to bring awareness to one's experiences without judgment. This technique includes the following steps: Stop or Slow down. Observe what is happening. Bring attention to Breathing. Expand awareness to the whole body. Respond mindfully, with awareness.

ELIGIBILITY:
Inclusion Criteria:

* Present for an intake appointment at study site for treatment of opioid use disorder.
* Eligible for receipt of buprenorphine-naloxone treatment (e.g. Suboxone, Bunavil, Zubsolv) as determined by clinic physicians
* 18 years or older
* Willing to be randomized to one of the two intervention arms
* Ability to comprehend consent and intervention materials (approximately 8th-grade level).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen J Derefinko, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Brief Motivational Intervention + Substance Free Activities + Mindfulness-Based Adherence Promotion: BSM (Brief Motivational Intervention + Substance Free Activities Session + Mindfulness-Based Adherence Promotion) participants had one-on-one behavioral intervention sessions at each of the first four visits after initiation of Buprenorphine-Naloxone.
Period: Overall Study
Arm/Group | Contingency management (CM) | Brief Motivational Intervention + Substance Free Activities + Mindfulness-Based Adherence Promotion
Started | 24 | 24
Completed | 22 | 22
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: 48 participants were randomized, but 4 never completed baseline/demographics assessments leaving N=44 with 22 in each arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Contingency Management (CM) | Brief Motivational Intervention + Substance Free Activities + Mindfulness-Based Adherence Promotion | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.45 (10.75) | 35.41 (9.88) | 37.43 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 20 | 22 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 14 | 13 | 27
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment Adherence
Description: Defined as no negative buprenorphine urine tests and attendance of at least two visits.
Time Frame: Through study completion, an average of 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Contingency management (CM) | Brief Motivational Intervention + Substance Free Activities + Mindfulness-Based Adherence Promotion
Number analyzed (Participants) | 22 | 22
Participants | 16 | 13

ADVERSE EVENTS:
Time Frame: Participants were systematically assessed for adverse events throughout their participation in the study which lasted for 6 months from baseline.
Description: Clinicaltrials.gov definitions were used.
Arm/Group | Contingency management (CM) | Brief Motivational Intervention + Substance Free Activities + Mindfulness-Based Adherence Promotion
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/22 | 1/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contingency management (CM) (N=22) | Brief Motivational Intervention + Substance Free Activities + Mindfulness-Based Adherence Promotion (N=22)
Incomplete spinal fusion (Surgical and medical procedures) | 0 (0) | 1 (1)
Overdose (Social circumstances) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT04464421/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT04464421/SAP_001.pdf
  • Informed Consent Form (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT04464421/ICF_002.pdf